CLINICAL TRIAL: NCT07299448
Title: Biological Determinants and Neural Compensatory Mechanisms of Oropharyngeal Dysphagia in Parkinson's Disease
Brief Title: Biological Determinants and Neural Compensation of Dysphagia in Parkinson's Disease
Status: Recruiting | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-2374; 529859742 (Other Grant/Funding Number: Deutsche Forschungsgemeinschaft (DFG))
Record Dates: First submitted 2025-11-26; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-09

CONDITIONS: Parkinsons Disease (PD); Oropharyngeal Dysphagia
Keywords: Dysphagia, Swallowing Disorder, Parkinson's Disease, Swallowing Compensation, Neuroimaging Biomarkers, Functional MRI, Proteomics
MeSH Terms: conditions — Parkinson Disease; Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and cerebrospinal fluid (CSF) samples will be retained for proteomic analyses. No DNA or genetic testing will be performed. Samples will be stored under standardized biobanking conditions for future protein-based investigations related to dysphagia and Parkinson's disease
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parkinson's Disease Patients with Dysphagia: Participants who have been diagnosed with Parkinson's disease and are still able to eat and drink independently. These individuals undergo a detailed examination of their swallowing function, compensatory mechanisms, and the neural correlates of dysphagia.

SUMMARY:
Parkinson's disease (PD) is the second most common neurodegenerative disorder and frequently leads to oropharyngeal dysphagia, a swallowing disorder that strongly affects patient health and quality of life. Dysphagia in PD is associated with aspiration pneumonia, malnutrition, and impaired medication intake, which together represent one of the leading causes of morbidity and premature mortality in these patients. Despite its clinical relevance, the underlying biological mechanisms of dysphagia in PD are not fully understood, and current treatment strategies are limited.

The purpose of this study is to investigate the clinical, biological, and neural determinants of oropharyngeal dysphagia in patients with PD, and to explore compensatory mechanisms of the brain that may counteract swallowing difficulties. We hypothesize that dysphagia in PD is linked not only to disease severity and progression but also to specific biological markers and neural plasticity in the swallowing network.

This is a prospective, cross-sectional observational study including 100 patients with PD. Swallowing function will be systematically assessed using flexible endoscopic evaluation of swallowing (FEES), a gold standard method for detecting penetration and aspiration. Additional clinical data will be collected, including motor and non-motor symptoms, disease severity, and quality of life measures. Biological assessments will include blood-based biomarkers related to inflammation and neurodegeneration. Furthermore, functional magnetic resonance imaging (fMRI) will be used to examine cortical and subcortical activity patterns associated with swallowing and to identify potential compensatory activation in dysphagic and non-dysphagic patients.

By integrating clinical, biological, and imaging approaches, this study aims to provide a comprehensive characterization of dysphagia in PD. The findings are expected to improve the understanding of disease mechanisms and to identify predictors of dysphagia onset and severity. Ultimately, this knowledge may help to guide the development of targeted therapeutic strategies, reduce the risk of severe complications, and improve quality of life for patients with Parkinson's disease.

DETAILED DESCRIPTION:
Background and Rationale Parkinson's disease (PD) is the second most common neurodegenerative disorder worldwide and is characterized by progressive motor and non-motor symptoms. Among its complications, oropharyngeal dysphagia (OD) is one of the most clinically relevant. Up to 80% of patients develop swallowing impairment during the course of the disease, often without recognizing its presence. Dysphagia is associated with aspiration pneumonia, malnutrition, dehydration, and impaired medication intake, representing a leading cause of morbidity and premature mortality in PD. Despite its high prevalence and impact, the underlying mechanisms of PD-related dysphagia are not fully understood, and current treatment options are limited.

Dysphagia in PD appears to be caused by a combination of central and peripheral factors. On the central level, dopamine deficiency contributes to motor dysfunction, including bradykinesia or freezing of swallowing. Cortical involvement and impaired sensorimotor integration may further reduce swallowing efficiency. On the peripheral level, impaired pharyngeal sensory function and reduced secretion of Substance P have been linked to silent aspiration and insufficient protective reflexes. Evidence from aging research and initial PD studies suggests that compensatory neural activity in cortical swallowing networks may mitigate the risk of aspiration in some patients. However, the clinical, biological, and neural determinants of preserved swallowing function and compensation in PD remain poorly defined.

Objectives and Hypotheses

The overarching objective of this study is to identify biological determinants and neural compensatory mechanisms of oropharyngeal dysphagia in PD. The specific aims are:

To characterize the prevalence, severity, and clinical phenotype of dysphagia in PD using standardized instrumental diagnostics.

To investigate biological determinants of swallowing impairment, including inflammatory and neurodegenerative markers in blood and saliva, sensory function, and proteomic signatures.

To examine neural correlates of swallowing function using task-based and resting-state functional magnetic resonance imaging (fMRI), diffusion tensor imaging (DTI), and muscle volumetry.

To identify clinical and biological factors associated with preserved neural compensation in PD, which may serve as potential therapeutic targets.

We hypothesize that dysphagia in PD is linked not only to disease progression but also to distinct biological markers and altered neural activity patterns. We further hypothesize that compensatory neural activation can be demonstrated in patients with mild dysphagia and that these mechanisms are modulated by clinical and biological determinants.

Study Design This is a prospective, cross-sectional observational study conducted at Heinrich-Heine-University Düsseldorf. A total of 100 patients with idiopathic PD across different disease stages will be recruited. The inclusion criterion is the ability to eat and drink orally and comply with study procedures. Exclusion criteria are tube feeding, other neurological or structural causes of dysphagia, severe comorbidities, or contraindications to MRI.

All participants will undergo a standardized study protocol consisting of three examination blocks:

Clinical and Instrumental Swallowing Assessment Swallowing will be assessed using Flexible Endoscopic Evaluation of Swallowing (FEES), which is considered a gold standard for detecting penetration, aspiration, and pharyngeal residue. The FEES protocol will include assessment of secretion management, swallowing of different consistencies, medication swallowing, dual-task swallowing (cognitive and motor load), pharyngeal sensitivity testing, and reflexive cough testing. Dysphagia severity and phenotype will be classified using validated scales.

Clinical, Biological, and Functional Assessments Clinical data will include demographics, disease duration, Hoehn & Yahr staging, motor severity (UPDRS), non-motor symptoms, cognitive testing, frailty, sarcopenia, nutritional status, hydration, immunosenescence, and quality of life measures. Biological samples (saliva and blood) will be collected for biomarker analysis, including Substance P, inflammatory cytokines, and proteomic profiling. Smell and taste testing will be performed to assess sensory function.

Neuroimaging All participants will undergo MRI scanning, including structural MRI, diffusion tensor imaging, muscle volumetry, and functional MRI during swallowing and sensory stimulation tasks. Task-based fMRI will examine cortical and subcortical swallowing networks, dual-task swallowing under cognitive or motor load, and pharyngeal sensory stimulation. Resting-state fMRI will be used to investigate functional connectivity. DTI will assess white matter integrity in swallowing-related pathways.

Outcome Measures The primary outcome is the presence and severity of dysphagia as determined by FEES.

Secondary outcomes include:

Biological markers associated with dysphagia severity. fMRI activation patterns reflecting neural compensation. Relationships between clinical phenotype, biomarkers, and imaging findings. Identification of predictors of preserved swallowing function.

Expected Impact This study will provide a comprehensive, multimodal characterization of oropharyngeal dysphagia in PD by integrating clinical, biological, and neuroimaging data. It will improve the understanding of disease mechanisms, identify predictors of dysphagia onset and severity, and shed light on neural compensatory mechanisms. Ultimately, the findings are expected to guide the development of targeted therapeutic strategies, support earlier diagnosis, and improve patient care. In the long term, the study may contribute to reducing complications such as aspiration pneumonia and malnutrition, improving quality of life, and lowering the healthcare burden associated with PD-related dysphagia.

ELIGIBILITY:
Inclusion Criteria:

.- Patients with idiopathic Parkinson's disease diagnosed according to the MDS diagnostic criteria

* Participation possible in all disease stages, regardless of the presence or absence of subjective or objective oropharyngeal dysphagia
* Cognitive ability sufficient to comply with the study paradigm
* Daily oral intake of food and fluids (exclusion of patients with exclusive tube feeding)

Exclusion Criteria:

* Presence of other conditions associated with oropharyngeal dysphagia, such as stroke, head and neck cancer, neuroinflammatory diseases, neuromuscular disorders, or other brain injuries
* Presence of electronic stimulation devices (e.g., pacemaker, deep brain stimulation) or other contraindications for MRI imaging
* Diagnosis of asthma or COPD (due to performance of the cough reflex test in "Block 1: Assessment of OD and pharyngeal hyposensitivity")

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients diagnosed with idiopathic Parkinson's disease according to the MDS diagnostic criteria (Postuma et al., 2015). Participants may be included in any stage of the disease, provided they are cognitively able to follow the study paradigm and are able to take food and liquids orally. Patients with exclusive tube feeding, comorbid conditions associated with oropharyngeal dysphagia (e.g., stroke, head and neck cancer, neuromuscular disorders), contraindications for MRI, or chronic pulmonary diseases such as asthma or COPD are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Dysphagia Severity assessed by Dynamic Imaging Grade of Swallowing Toxicity-Fiberoptic Endoscopic Evaluation of Swallowing (DIGEST-FEES) | Baseline
  Swallowing safety and efficiency will be assessed using the Dynamic Imaging Grade of Swallowing Toxicity-Fiberoptic Endoscopic Evaluation of Swallowing (DIGEST-FEES). The DIGEST-FEES is a validated, ordinal rating scale that integrates measures of airway invasion (penetration-aspiration) and pharyngeal residue to generate a composite severity grade of dysphagia. Scores range from 0 (no dysphagia) to 4 (life-threatening dysphagia), with higher scores indicating greater swallowing impairment.

SECONDARY OUTCOMES:
Neural Activation Patterns (fMRI) | Baseline
  Functional brain activity during swallowing tasks will be assessed using fMRI. Focus is on compensatory activation patterns in cortical and subcortical areas associated with swallowing control.
Electromyography (EMG) of Swallowing Muscles | Baseline
  Surface EMG recordings will assess the number of swallows during fMRI
Change in Global Cognitive Function as Assessed by the Montreal Cognitive Assessment (MoCA) | Baseline
  Global cognitive function will be assessed using the Montreal Cognitive Assessment (MoCA), a validated, brief screening tool designed to detect mild cognitive impairment and broader cognitive dysfunction. The MoCA evaluates multiple cognitive domains, including:
  Attention and concentration
  Executive functioning
  Memory
  Language
  Visuospatial skills
  Abstraction
  Orientation
  Total scores range from 0 to 30, with higher scores indicating better cognitive performance. A change in MoCA score over time will be used to assess change in overall cognitive function.
Change in Swallowing-Related Quality of Life as Assessed by the Swallowing Quality of Life Questionnaire (SWAL-QOL) | Baseline
  Swallowing-related quality of life will be assessed using the Swallowing Quality of Life Questionnaire (SWAL-QOL), a validated, patient-reported outcome measure designed specifically to evaluate the impact of dysphagia on daily functioning and well-being. The SWAL-QOL consists of 44 items across multiple domains, including:
  Burden
  Eating duration
  Eating desire
  Food selection
  Communication
  Fear
  Mental health
  Social functioning
  Fatigue
  Sleep
  Item responses are converted to domain and total scores typically scaled from 0 to 100, with higher scores indicating better swallowing-related quality of life. Change in SWAL-QOL total score (and/or domain scores) over time will be used to assess patient-perceived treatment effect.
Change in Airway Invasion Severity as Assessed by the Penetration-Aspiration Scale (PAS) | Baseline
  Airway invasion during swallowing will be assessed using the Penetration-Aspiration Scale (PAS), an 8-point, validated, ordinal scale that quantifies the depth of bolus entry into the airway and the individual's response to that invasion during instrumental swallowing assessment. Scores range from 1 to 8, where:
  1 = Material does not enter the airway
  2-5 = Penetration (material enters the airway but remains above the vocal folds)
  6-8 = Aspiration (material passes below the vocal folds), with higher scores indicating more severe impairment and reduced protective response
  Higher PAS scores indicate greater severity of airway compromise and increased aspiration risk.
Change in Pharyngeal Residue Severity as Assessed by the Yale Residue Severity Scale (YRSS) | Baseline
  Pharyngeal residue following swallowing will be assessed using the Yale Residue Severity Scale (YRSS), a validated, ordinal rating scale designed for use with Fiberoptic Endoscopic Evaluation of Swallowing (FEES). The YRSS quantifies the amount of post-swallow residue within two key anatomical locations:
  Valleculae
  Pyriform sinuses
  Each site is scored separately on a 5-point scale:
  0 = No residue
  1. = Trace residue
  2. = Mild residue
  3. = Moderate residue
  4. = Severe residue (nearly full or full pooling)
  Higher scores indicate greater impairment in swallowing efficiency and increased risk for post-swallow airway invasion.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Düsseldorf, Düsseldorf, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Yes
demographic data, clinical description of the cohort, and results of the examinations
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: beginning of recruitment until end of study